CLINICAL TRIAL: NCT05100901
Title: Tolerance and Safety of an Oral Nutritional Supplement Containing Monoacylglycerol Oil (MAG Oil) as the Main Lipid Source in Healthy Adolescents and Adults
Brief Title: Tolerance and Safety of an Oral Nutritional Supplement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Adolescent cohort will be conducted as separate trial
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2104CLI
Record Dates: First submitted 2021-08-16; First posted 2021-10-29 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2022-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral nutritional supplement (Experimental): Oral nutritional supplement that contains MAG oil
  Interventions: Dietary Supplement: MAG oil oral nutritional supplement (ONS)

INTERVENTIONS:
Dietary Supplement: MAG oil oral nutritional supplement (ONS) — The study product is suitable for use as an oral nutritional supplement (ONS).The study product contains MAG oil, hydrolyzed whey protein, simple carbohydrates, vitamins and minerals.

SUMMARY:
This is an open label, non-randomized, interventional, single arm study.

DETAILED DESCRIPTION:
Primary objective is to assess whether the MAG oil (monoacylglycerol oil) containing study formula is well tolerated and safe when used as an ONS in healthy adults and adolescents.

Secondary objectives:

1. Describe the incidence and characteristics of possible gastrointestinal intolerance symptoms
2. Describe changes in stool characteristics, specifically stool frequency and consistency
3. Describe changes in anthropometric parameters, particularly weight and body mass index (BMI)
4. Describe changes in blood parameters of lipid metabolism
5. Describe changes in hematological and serum biochemistry parameters
6. Describe daily ONS intake and assess dietary adherence to the study protocol

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* BMI range from >18 to <28 kg/m2 for adults with a minimum body weight of 45 kg
* BMI range between the 25th and 90th percentile according to the Swiss growth charts for adolescents with a minimum body weight of 40 kg
* Cohort 1: Adults aged 18+ years (6 males, 6 females)
* Cohort 2: Adolescents aged 12-17 years (6 males, 6 females)
* Deemed able to comply with study protocol for 2 weeks
* Able to obtain written informed consent from participants and /or legal guardians

Exclusion Criteria:

* Pre-existing chronic medical or psychiatric conditions, as diagnosed by the treating physician
* Subjects taking dietary supplements (energy supplements, protein supplements) will be excluded. Subjects can continue taking vitamin or herbal supplements during the study period.
* Abnormal bowel transit, history of a gastrointestinal disorder (e.g., inflammatory bowel disease (IBD), diverticular disease, colon cancer, irritable bowel syndrome (IBS), history of chronic constipation with passage of fewer than 3 spontaneous bowel movements per week on average, or chronic or recurrent diarrhea with loose or watery bowel movements more than 3 times daily.
* Recent episode of an acute gastrointestinal illness with significant gastrointestinal symptoms in the 7 days prior to enrolment.
* Colonoscopy or other bowel cleansing procedures within 4 weeks prior to enrolment.
* Prior use of prescription medication(s), in particular antibiotics, antacids, laxatives or other medications impacting gastrointestinal transit time, within 8 weeks prior to enrolment.
* Significant medical or surgical event in the past 3 months potentially interfering with study procedures and assessments.
* Known food allergy in particular cow's milk protein allergy (CMPA) or known hypersensitivity/intolerance to any other ingredients in the study product.
* Known alcohol or substance abuse; specifically, alcohol intake > 2 servings per day. A serving is 0.4 dl of strong alcohols, 1 dl of red or white wine, or 3 dl of beer.
* Pregnant or lactating women or having given birth in the past 6 months prior to enrolment.
* Family or hierarchical relationships with Clinical Innovation Lab staff.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Number of subjects who develop gastrointestinal intolerance leading to premature discontinuation | [ Time Frame: Day 2 to Day 15 ]
  Number of subjects who develop gastrointestinal intolerance reported as adverse events related to the investigational product and leading to premature discontinuation of the study product, assessed by a daily questionnaire

SECONDARY OUTCOMES:
Severity of gastrointestinal intolerance symptoms | [ Time Frame: Day 2 to Day 14 ]
  Visual analog scale from 0 (no symptom) to 10 (maximum severity)
Severity of gastrointestinal intolerance symptoms | [ Time Frame: Day 1 and Day 15 ]
  Gastrointestinal Symptom Rating Scale, each visit will asses symptoms over the past 7 days
Change in stool frequency | [ Time Frame: Day 1 to Day 15 ]
  Assessed by a questionnaire for stool frequency
Change in weight | [ Time Frame: Day 1 and Day 15 ]
Change in triglycerides | [ Time Frame: Day 1 and Day 15 ]
Change in cholesterol | [ Time Frame: Day 1 and Day 15 ]
Change in fatty acids profile | [ Time Frame: Day 1 and Day 15 ]
Changes full blood count | [ Time Frame: Day 1 and Day 15 ]
  Number of participants with changes in haematology measurements (erythrocyte count, thrombocyte count, haemoglobin, haematocrit, mean cell hemoglobin concertation) using immunoassays.
Changes liver function | [ Time Frame: Day 1 and Day 15 ]
  Number of participants with changes in liver function measurements (AST, ALT, ALP, GGT, albumin) using immunoassays
Changes in renal function | [ Time Frame: Day 1 and Day 15 ]
  Number of participants with changes in renal function measurements (urea, creatinine) using immunoassays
Changes in blood glucose | [ Time Frame: Day 1 and Day 15 ]
Daily intake of study product | [ Time Frame: Day 1 to Day 15 ]
  Number of subjects adhering to daily intake of the study product from baseline to Day 15, assessed by a daily questionnaire
Change in stool consistency | [ Time Frame: Day 1 to Day 15 ]
  Assessed by the Bristol Stool Scale
Change in BMI | [ Time Frame: Day 1 and Day 15 ]
Change in Fat soluble-vitamins profile | [ Time Frame: Day 1 and Day 15 ]
  Fat soluble-vitamins (A, D, E, K)
Change in serum biochemistry parameters | [ Time Frame: Day 1 and Day 15 ]
  Number of participants with changes in serum biochemistry (triglycerides, total protein, bilirubin total, bilirubin direct, sodium, potassium, calcium, phosphate, magnesium, chloride, CRP) using immunoassays

CONTACTS AND LOCATIONS:
Locations (1):
- Nestlé CDU / Clinical Innovation Lab, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zemrani B, Krattinger LF, Giuffrida F, Corthesy J, Ran-Ressler RR, Benyacoub J. Safety and tolerability of Monoacylglycerol-rich oil as a novel predigested dietary fat source of an enteral formula in healthy adults and adolescents: Two single-arm, open-label studies. Clin Nutr ESPEN. 2025 Feb;65:339-347. doi: 10.1016/j.clnesp.2024.12.014. Epub 2024 Dec 15. PMID 39681164